CLINICAL TRIAL: NCT02656615
Title: An Open Label Biomarker Driven Phase II Clinical Trial of Abiraterone Acetate (AA) Re-Challenge in Patients With Metastatic Castration-Resistant Prostate Cancer and Prior Response to AA
Brief Title: Abiraterone-Rechallenge Study for CRPC Patients
Acronym: ABI-RE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of Patient accrual
Sponsor: Aurelius Omlin (Other)
Collaborators: Cantonal Hospital of St. Gallen (Other); University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor-Investigator, Aurelius Omlin, MD, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTU 14/020
Record Dates: First submitted 2016-01-04; First posted 2016-01-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abiraterone (Experimental): Abiraterone acetate 1000 mg once daily and Prednisone 2x5 mg daily (continuously as per prescription label).
  Interventions: Drug: abiraterone acetate

INTERVENTIONS:
Drug: abiraterone acetate — Abiraterone acetate 1000 mg once daily and Prednisone 2x5 mg daily (continuously as per prescription label).
  Other Names: Zytiga

SUMMARY:
To assess activity of abiraterone-re-challenge in patients with advanced prostate cancer and prior response to abiraterone.

DETAILED DESCRIPTION:
To assess activity of abiraterone-re-challenge in patients with advanced prostate cancer and prior response to abiraterone. CRPC patients with prior response to abiraterone (confirmed PSA Response) and progression can be re-challenged with abiraterone. Patients may have received treatment with docetaxel, enzalutamide and radium-223.

ELIGIBILITY:
Inclusion Criteria:

1. Written prostate cancer.
2. Adult patients with histological or cytological diagnosis of adenocarcinoma of the prostate.
3. Men with castration-resistant metastatic decline maintained for at least 3 weeks as per PCWG2 criteria).
4. Confirmed biochemical response to prior abiraterone acetate (≥50% PSA Informed Consent (including consent for biomarker studies including the fresh tumour biopsies)
5. Progressive disease according to PCWG2 criteria during prior therapy with standard dose of abiraterone acetate (confirmed increase of PSA ≥25% over nadir) or soft-tissue or bone progression. Patients that have stopped abiraterone acetate for reasons other than progression are not eligible.
6. Documented progression of disease by any of the criteria listed here:

   * PSA
   * Soft tissue
   * Bone scan all as per PCWG2 criteria
7. Patients may have received treatment with docetaxel, enzalutamide or radium-223
8. PSA of ≥10ug/l
9. ECOG performance status 0 - 2
10. At least 3 months (90 days) since stop of prior abiraterone acetate.

Exclusion Criteria:

1. Major surgery within 28 days weeks prior to start of treatment
2. Prior treatment with cabazitaxel or the CYP-17 inhibitor TAK-700/orteronel
3. Any concurrent treatment or prior treatment with an investigational drug within 28 days prior to start of treatment.
4. Known brain or leptomeningeal disease
5. Concurrent use of steroids other than prednisone >10mg/d
6. Inadequate bone marrow and organ function as evidenced by:

   Platelet count <75 x 10 G/L ASAT and/or ALAT ≥ 2.5 x ULN Total bilirubin ≥ 1.5 x ULN (≥ 2.0 x ULN for patients with Gilbert's disease) Hypokalaemia despite adequate supplementation Creatinine Clearance <30ml/min
7. Uncontrolled hypertension or cardiac failure or LVEF <50%

creatinine clearance is to be calculated by using the formula of Cockcroft-Gault in appendix 4 of the protocol

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Response rate | at week 12
  Soft-tissue and PSA Response per PCWG2

SECONDARY OUTCOMES:
Rate of CTC conversion | Measured at baseline and at 12 weeks
  Rate of CTC conversion from a baseline count of ≥5/7.5ml to <5/7.5ml
Rate of PSA decline 30% | at week 12
  Rate of PSA declines of ≥30% at 12 weeks and at any time on study thereafter
rPFS | From date of start of treatment up to 6 months
  From date of start of treatment until the date of first documented progression or date of death from any cause, whichever came first
Disease control rate | at 12 and 24 weeks
  Disease control rate at 12 and 24 weeks (defined as SD, PR, CR, see response criteria)

CONTACTS AND LOCATIONS:
Overall Officials: Aurelius G Omlin, MD, Principal Investigator — Cantonal Hospital of St. Gallen
Locations (3):
- Switzerland (3):
  - Cantonal Hospital Chur, Chur, Kanton Graubünden
  - University Hospital Basel, Basel
  - Cantonal Hospital St.Gallen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No